CLINICAL TRIAL: NCT03084874
Title: Efficacy of a Coaching Program to Promote Physical Activity and Reduce Sedentary Behavior After a COPD Exacerbation That Require Hospitalization
Brief Title: Efficacy of a Coaching Program to Promote Physical Activity and Reduce Sedentary Behavior After a COPD Hospitalization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Spanish Society of Pneumology and Thoracic Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR(AG)390/2015
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Physical Activity; Sedentary Lifestyle
Keywords: COPD; Physical Activity; Sedentary behaviour; Hospitalization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will receive an individualized coaching program to increase physical activity and reduce sedentary behavior during 12 weeks
  Interventions: Behavioral: Physical activity and sedentary behavior coaching program
- Control group (No Intervention): Patients in the control group will receive the standard care for patients with COPD during 12 weeks.

INTERVENTIONS:
Behavioral: Physical activity and sedentary behavior coaching program — The intervention group will receive an individualized coaching program. During a motivational interview an experienced physiotherapist will asses participant's usual exercise habits, possible barriers and facilitators, self-efficacy and motivation to increase physical activity and reduce sedentary time. Based on these data (and baseline physical activity/sedentary information) an individualized, progressive program with specific goals setting and self-monitoring will be established (patients will be active participants and decision makers in this process).
  Arms: Intervention group

SUMMARY:
Patients with COPD are more inactive and more sedentary than subjects of the same age and patients with other chronic diseases. This inactivity and sedentary behavior is accentuated after hospitalizations due to a COPD exacerbation, and it increases the risk for future hospitalizations and mortality. Therefore, there is a need for intervention to promote physical activity and to reduce sedentary behavior after these events. The present study aims to evaluate the efficacy of a coaching program to promote physical activity and reduce sedentary behavior in patients with COPD who have suffered a hospitalization due to a COPD exacerbation. Sixty-six COPD patients admitted to the hospital will be recruited during 18 months. Physical activity, sedentary behaviors, as well as other clinical and functional parameters will be evaluated after hospital discharge. Patients will be then randomized to an intervention and control group (1:1). The intervention group will receive an individualized coaching program. During a motivational interview an experienced physiotherapist will asses participant's usual exercise habits, possible barriers and facilitators, self-efficacy and motivation to increase physical activity and reduce sedentary time. Based on these data (and baseline physical activity/sedentary information) an individualized, progressive program with specific goals setting and self-monitoring will be established (patients will be active participants and decision makers in this process). The control group will receive the usual care during follow-up. Physical activity, sedentary behaviors, as well as the clinical and functional variables will be evaluated again at 12 weeks in both patients' groups.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of COPD according to spirometric criteria (post-bronchodilator FEV1 / FVC less than 70%)
2. Smoking exposure> 10 paq/year.
3. Age greater than 40 years.
4. Hospitalization due to a COPD exacerbation
5. Written informed consent.

Exclusion Criteria:

1. Patients needing the care of an Intensive Care Unit.
2. Patients who have been hospitalized more than once for a COPD exacerbation in the previous 12 months (at least 3 months from last discharge).
3. Patients with continuous oxygen therapy who do not have a portable source before admission.
4. Patients with severe hypoxemia at rest (SpO2 <85% at rest) at discharge
5. Mental incapacity, severe comorbidity, general fragility or advanced age that could substantially difficult patient's participation in the study.
6. Patients who need mechanical aids for walking.
7. Patients participating in a pulmonary rehabilitation program.
8. Difficulty understanding Spanish / Catalan.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in steps per day | Baseline and 12 weeks
  Steps per day will be objectively measured with an accelerometer
Change in the number of active periods per day | Baseline and 12 weeks
  Number of periods spent standing, walking or shuffling objectively measured with an accelerometer
Change in time spend in light and moderate physical activity | Baseline and 12 weeks
  Time spend in light and moderate physical activity (1.5-3 and 3-6 METS) objectively measured with an accelerometer
Change in time spend in sedentary behavior | Baseline and 12 weeks
  Time spend in sedentary behavior (sitting or lying) objectively measured with an accelerometer
Breaks in sedentary behaviour | Baseline and 12 weeks
  Number of transitions from sedentary behavior to standing or walking objectively measured with an accelerometer

SECONDARY OUTCOMES:
Change in exercise capacity | Baseline and 12 weeks
  Distance walked in the 6-minute walk test
Change in muscle force | Baseline and 12 weeks
  Quadriceps muscle force tested with a hand-held dynamometer
Change in patient's quality of life | Baseline and 12 weeks
  patient's quality of life measured using the St. George's Respiratory Questionnaire (SGRQ) anbd the COPD assesment test (CAT)

OTHER OUTCOMES:
Change in patients's anxiety and depression | Baseline and 12 weeks
  Patient's anxiety and depression measured using the Hospital Anxiety and Depression scale (HADS)
Change in dyspnoea during daily activities | Baseline and 12 weeks
  Dyspnoea during daily activities measures using the London Chest Activity of Daily Living scale (LCADL)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared